CLINICAL TRIAL: NCT02360163
Title: The "Peripheral Access Utilizing Sonographic Evaluation" Study
Acronym: PAUSE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No enrollment was achieved
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro 2921
Record Dates: First submitted 2015-02-05; First posted 2015-02-10 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: DIVA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Landmark Technique Attempt (Active Comparator): Patients will undergo an additonal TLT attempt
  Interventions: Procedure: Traditional Landmark Technique (TLT)
- USGPIVA Technique Attempt (Experimental): Patients will be offered a USGPIVA attempt after two failed attempts using the traditional landmark technique (TLT)
  Interventions: Device: ultrasound guided peripheral intravenous access (USGPIVA)

INTERVENTIONS:
Procedure: Traditional Landmark Technique (TLT)
  Arms: Landmark Technique Attempt
Device: ultrasound guided peripheral intravenous access (USGPIVA)
  Arms: USGPIVA Technique Attempt

SUMMARY:
The purpose of this study is to reduce, by using the ultrasound guided technique, the minor surgical procedures that might be required to deliver fluids into the blood of critically ill patients simply because the patients' veins cannot be located through the manual technique.

DETAILED DESCRIPTION:
The purpose of this study is to reduce, by using the ultrasound guided technique, the minor surgical procedures that might be required to deliver fluids into the blood of critically ill patients simply because the patients' veins cannot be located through the manual technique.

The ultrasound assisted technique will increase accessibility to small veins that might be missed via the manual technique. The technique of using an ultrasound machine to assist the administration of fluids into a patient's veins is called ultrasound guided peripheral intravenous access (USGPIVA), while the traditional technique that uses only sight and touch to locate a patient veins without machine assistance is called the traditional landmark technique (TLT). The investigators will compare the effectiveness of USGPIVA with TLT in terms of reducing complications and costs.

ELIGIBILITY:
Inclusion Criteria:

* The patient is >= 21 years of age
* Adult critically ill patients in CCU and MICU requiring short peripheral intravenous access
* The patient has been identified as difficult intravenous access (DIVA), defined as at least two failed blind sticks in the antecubital fossa or more distal upper arm veins
* The patient does not otherwise require a CVC

Exclusion Criteria:

* The patient has a PICC line on the same side as IV placement and has the following:

  * Has a condition poses risk for DIC, inadequate flow, or infection.
  * Has been identified as a site for "Save the Vein" protocol implementation, unless permission is otherwise obtained by the patient's physician.
  * Has a hemodialysis fistula in place on that upper arm side.
* The patient is expected to require therapeutic agent or procedure that necessitates central venous access such as:

  * central venous monitoring
  * Total Parenteral Nutrition
  * Antibiotic requiring central venous access
  * Chemotherapy
  * Vesicants
  * Medications pH less than 5 or more than 9
  * Medications of glucose concentrations above 10%
  * Solution with protein concentrations above 5% (Vascular Access Management, n.d.)
* The patient already has a central venous catheter access, for reasons other than DIVA, through which therapy can be infused
* The patient has renal disease and a "Save The Vein" order is anticipated or pending (serum creatinine >2mg/dL and GFR <20) for one of the patient's arms, unless permission is otherwise obtained by the patient's physician
* The patient has a bleeding disorder, unless permission is otherwise obtained by the patient's physician
* The clinician believes the patient is not a good fit for the study or that the procedure is not appropriate for patient at the given moment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2017-01-19 (Actual); Study Completion 2017-01-19 (Actual)

PRIMARY OUTCOMES:
Reduction in number of minor surgical procedures that may be required to deliver fluids into the blood of critically ill patients by using the ultrasound guided technique | 1 Day

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Van Buitenen, MSN, APN, RN, Principal Investigator — Hackensack UMC
Locations (1):
- Hackensack University Medical center, Hackensack, New Jersey, United States

REFERENCES:
- [Derived] Tada M, Yamada N, Matsumoto T, Takeda C, Furukawa TA, Watanabe N. Ultrasound guidance versus landmark method for peripheral venous cannulation in adults. Cochrane Database Syst Rev. 2022 Dec 12;12(12):CD013434. doi: 10.1002/14651858.CD013434.pub2. PMID 36507736